CLINICAL TRIAL: NCT06397651
Title: A Decentralized, Double-blinded, Randomized, 18 Month, Parallel-group, Superiority Study to Evaluate the Impact of Complement Theory's Live Coactive Exercise Coaching and Personalized Digital Application on Cancer Survivors' Quality of Life
Brief Title: A Randomised Controlled Trial to Evaluate the Impact of Complement Theory's Live CoActive Exercise Coaching and Personalized Digital Application on Cancer Survivors' Quality of Life
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Complement Theory Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Pro00077693
Record Dates: First submitted 2024-04-25; First posted 2024-05-03 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Lung Cancer; Prostate Cancer; Colorectal Cancer; Other Cancer
Keywords: Other cancer here refers to all cancers apart from Breast, Lung, Prostate and Colorectal Cancer
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Treatment Group
  * Participants will get access to Complement Theory's Live Coaching program, focusing on Exercise and Meditation and supplemented with evidence-based information on Diet, Sleep, and other lifestyle practices, adjunct to the core treatment.
  * Each week, up to five sessions of 45 minutes each will be offered, with a recommendation for participants to engage in a minimum of 3 sessions.
  * Each session will consist of 30 Minutes of Physical Exercise and 7 minutes of meditation. Each session will be a combination session focused on Aerobic and Strength, with flexibility and balance exercises included as supplements.
  Active Comparator (Control) Group
  * Participants in this group will receive access to a curated collection of publicly available guidelines for lifestyle modification. These resources, presented through a digital application, will focus on exercise, meditation, diet, and sleep, but without the live coaching or program personalization.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Live CoActive Coaching program, focusing on Exercise and Meditation, along with evidence-based information on Diet, for 18 months
  Interventions: Behavioral: Complement Theory's Live CoActive Exercise Coaching and Personalized Digital Application
- Control Group (Active Comparator): 18 months access to Digital application with expert guidelines on lifestyle modification focusing on exercise, meditation, as well as information on diet, sleep and other lifestyle practices. Does not include live coaching and personalization.
  Interventions: Behavioral: Digital application with expert guidelines on lifestyle modification

INTERVENTIONS:
Behavioral: Complement Theory's Live CoActive Exercise Coaching and Personalized Digital Application — Participants will get access for 18 months to Complement Theory's Live CoActive Coaching program, focusing on Exercise and Meditation and supplemented with evidence-based information on Diet, adjunct to the core treatment.
  * Each week, up to five sessions of 45 minutes each will be offered, with a recommendation for participants to engage in a minimum of three sessions to ensure adequate program exposure and benefits.
  * Each session will consist of 30 Minutes of Physical Exercise and 7 minutes of meditation. Each session will be a combination session focused on Aerobic and Strength, with flexibility and balance exercises included as supplements.
  Arms: Test Group
Behavioral: Digital application with expert guidelines on lifestyle modification — 18 months access to Digital application with expert guidelines on lifestyle modification focusing on exercise, meditation, as well as information on diet, sleep and other lifestyle practices.
  Arms: Control Group

SUMMARY:
A Decentralized, Double-blinded, Randomized, 18 month, Parallel-group, Superiority Study to evaluate the impact of Complement Theory's Live Coactive Exercise Coaching and Personalized Digital Application on Cancer Survivors' Quality of Life

DETAILED DESCRIPTION:
The randomized controlled trial (RCT) aims to evaluate the efficacy of Complement Theory's (CT) personalized and interactive, evidence-backed lifestyle program in improving Cancer Survivors' Quality of Life across all major cancer types.

Distinct from conventional interventions, CT's program offers live CoActive coaching through a mobile app, concentrating on Exercise and Meditation, and is enriched with evidence-based advice on Diet. This trial is pivotal in assessing the program's effectiveness against an active comparator - expert-recommended lifestyle modification resources suitable for cancer survivors -- to isolate the impact of coaching and personalization.

The primary objective is to investigate whether CT's novel approach can significantly improve Quality of Life for survivors. Furthermore, the trial seeks to measure absenteeism and presenteeism at work to provide a holistic evaluation of the program's impact on patient care and well-being. As an exploratory effort, the trial will also measure changes in healthcare expenditure across all survivors along with assessing cancer progression, recurrence in Prostate, Lung and Colorectal cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Cancer Type: Breast, Prostate, Colorectal, Lung and Other Cancer
* Cancer Stage: Stage 1 to 4
* Treatment Status: Has undergone any cancer-related treatment in last 12 months
* Age: Above 21 years
* Permission to access to last 1 year digital health records
* Access to smartphone or a tablet

Exclusion Criteria:

* Excludes individuals who have undergone surgery within the last 4 weeks or will undergo surgery in the next 4 weeks
* Participants declared medically unfit by their physicians to do physical exercise
* ECOG Score 3,4 or 5

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2024-05-12 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Impact of the program cancer survivors' Quality of Life Scores (QoLS), measured by the FACT-G instrument. | 18 months
  To quantify the impact of Complement Theory's Program on cancer survivors' Quality of Life, as measured by the change in FACT-G scores over the course of the trial.

SECONDARY OUTCOMES:
Effect on Employee Absenteeism | 18 Months
  Quantify the effect of CT's program on employee absenteeism by tracking changes in the number of sick days taken by participants.
Impact on Employee Presenteeism | 18 Months
  Determine the program's impact on employee presenteeism by assessing changes in work motivation and employee performance review scores.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio L. Battaglini, PhD, Principal Investigator — University of North Carolina; Erik Hanson, PhD, Principal Investigator — University of North Carolina
Locations (1):
- Complement Theory Inc., Dover, Delaware, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data shall be shared. This includes both primary and secondary outcomes related data points.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available 3 months after the end trial and will be available for 2 years after the date of availability.
Access Criteria: Anyone shall be able access after following a simple data request process. The person has to detail the purpose and expected outcomes, which will be reviewed and approved by the Principal Investigators.
  Plus, we will also ensure appropriate documentation. We will employ a data use agreement to prohibit re-identification attempts and ensure data is used as per the agreed proposal.
  The overall process has been designed to make the data access as open as possible and as closed as necessary, to protect participant privacy and reduce the risk of data misuse.

DOCUMENTS (2):
  • Study Protocol (2025-08-26): https://cdn.clinicaltrials.gov/large-docs/51/NCT06397651/Prot_002.pdf
  • Informed Consent Form (2024-04-09): https://cdn.clinicaltrials.gov/large-docs/51/NCT06397651/ICF_001.pdf